CLINICAL TRIAL: NCT03025477
Title: Randomized Study Assessing Two Strategies of First Line: a Strategy With Intraperitoneal Chemotherapy and a Strategy With Total Intravenous Strategy, in Patients With Epithelial Advanced Ovarian Cancer
Brief Title: Two Therapeutic Strategies in First-line in Patients With Epithelial Advanced Ovarian Cancer
Acronym: CHIMOVIP
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Groupe Hospitalier Diaconesses Croix Saint-Simon (Other)
Collaborators: GERCOR - Multidisciplinary Oncology Cooperative Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RVT_2015_2
Record Dates: First submitted 2016-12-15; First posted 2017-01-19 (Estimated); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Ovarian Cancer, Epithelial
Keywords: Intraperitoneal; Intravenous; Completeness of cytoreduction score; Carboplatin; Epirubicin; Paclitaxel; Cisplatin
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial | interventions — Paclitaxel; Epirubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control arm (Active Comparator): Initial or interval surgery associated with 6 cycles of chemotherapy in intravenous (IV) of carboplatin and paclitaxel.
  The regimen of administration of the chemotherapy is as following:
  * Carboplatin AUC 6 - IV - Day (D) 1
  * Paclitaxel 80mg / m² - IV - D1, D8, D15
  one cycle every 3 weeks
  Interventions: Drug: CC0 - Carboplatin (IV) - Paclitaxel (IV); Drug: CC>0 - Carboplatin (IV)- Paclitaxel (IV)
- Experimental arm (Experimental): Initial or interval surgery associated with 6 cycles of chemotherapy of cisplatin and epirubicin.
  * Cisplatin is administrated in intraperitoneal (IP) if no macroscopic residual tumor at the end of the intervention (initial or interval). If evidence of macroscopic residual tumor, cisplatin is administered in IV. Epirubicin is always given in IV.
  * Second cytoreduction surgery at mid-term of chemotherapy cycles, only in patients operable in response after 3 cycles and with persistent residual disease after initial surgery or incomplete initial staging.
  The regimen of administration of the chemotherapy is as following:
  * Cisplatin 80mg / m² - IV or IP - D1
  * Epirubicin 60mg / m² - IV - D3
  one Cycle every 3 weeks.
  Interventions: Drug: CC0 - Cisplatin (IP) - Epirubicin (IV); Drug: CC>0 - Cisplatin (IP/IV)- Epirubicin (IV)

INTERVENTIONS:
Drug: CC0 - Carboplatin (IV) - Paclitaxel (IV) — (6 cycles)
  Arms: Control arm
Drug: CC0 - Cisplatin (IP) - Epirubicin (IV) — (6 cycles)
  Arms: Experimental arm
Drug: CC>0 - Carboplatin (IV)- Paclitaxel (IV) — * carboplatin (IV) - paclitaxel (IV) (3 cycles)
  * Interval surgery
  * Carboplatin (IV) - paclitaxel (IV) (3 cycles)
  Arms: Control arm
Drug: CC>0 - Cisplatin (IP/IV)- Epirubicin (IV) — * Cisplatin (IV) - Epirubicin (IV) (3 cycles)
  * Interval surgery :
    * if CC0: Cisplatin (IP) - Epirubicin (IV) (3 cycles)
    * if CC>0 Cisplatin (IV)- Epirubicin (IV) (3 cycles)
  Arms: Experimental arm

SUMMARY:
CHIMOVIP is a study to determine the best therapeutic strategy in patient with ovarian advanced cancer.

DETAILED DESCRIPTION:
This is a randomized phase II study, open-label and multicentric. After initial intervention (debulking surgery or diagnostic surgery) patient will randomized in the study according to Completeness of cytoreduction (CC) score (CC0 or CC>1).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed advanced (FIGO stage III or IV) invasive epithelial ovarian cancer, primary peritoneal cancer, or fallopian-tube cancer. Pleural cytology has to be performed in patients with pleural effusion.
* Initial intervention : debulking surgery or diagnostic surgery in the 3 weeks before inclusion
* Age ≥18 and < 75 years old.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 before surgery (ECOG ≤ 1 and Lee score < 6 in patients > 70 years old).
* Adequate blood count (test realized in the past 14 days before inclusion) : neutrophils > 1500/mm3, platelets > 150 000/mm3.
* Creatinine clearance MDRD ≥ 60 mL/min
* Registration in a national health care system (CMU included).
* Signed and dated informed consent.

Exclusion Criteria:

* FIGO stage IV extra-abdominal disease, with the exception of lymph nodes and pleural invasion.
* Patient having received previous chemotherapy for ovarian cancer.
* Left ventricular ejection fraction < 50% before chemotherapy initiation
* Other invasive cancer in the past 5 years (baso- and spinocellular cutaneous carcinoma with complete resection are accepted)
* Concomitant administration of prophylactic phenytoin or live attenuated viral vaccines such as yellow fever vaccine,
* Patients with known hypersensitivity to any component of study drug
* Patients without motivation or capacity to respect study requirements and constraints
* Pregnancy or breast feeding women

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2016-10 (Actual); Primary Completion 2021-10 (Estimated); Study Completion 2032-10 (Estimated)

PRIMARY OUTCOMES:
Pathological complete peritoneal response (pCR) | 2-year
  Interval debulking surgery or final evaluation peritoneal surgery

SECONDARY OUTCOMES:
Quality of life (QLQ -C30) assessment | Up to 2-year (at inclusion, after 3 cycles and end of treatment)
Quality of life (QLQ-OV28) assessment | Up to 2-year (at inclusion, after 3 cycles and end of treatment)
IPSS score | Up to 2-year (at inclusion, after 3 cycles and end of treatment)
Number of patients with treatment-related adverse events as assessed by CTCAE version 4.03 | 2-year
Event-free survival (EFS) | At 5-year and 10-year
Objective response rate at the various surgical step | Up to 2-year
Overall survival (OS) | At 5-year and 10-year

CONTACTS AND LOCATIONS:
Overall Officials: Richard VILLET, MD, Principal Investigator — Groupe Hospitalier Diaconessess Croix Saint Simon
Locations (7):
- France (7):
  - Centre Georges François Leclerc, Dijon
  - Institut Hospitalier Franco-Britannique, Levallois-Perret
  - Groupe Hospitalier Diaconesses Croix Saint Simon, Paris
  - Hôpital Saint Antoine, Paris
  - Hôpital Poissy Saint Germain, Poissy
  - CHU Poitiers, Poitiers
  - Centre Hospitalier Senlis, Senlis